## CLINICAL STUDY COVER PAGE

**Official Study Title:** Can Ultrasound-Guided Bilateral Cervical Plexus Block Combined With Translaryngeal Block For Tracheostomy Be An Alternative To General Anesthesia?

Namık Kemal University ethics committee with the protocol number: 2020.240.10.08

Namık Kemal University ethics committee approval date: October 27, 2020

Address for correspondence: Dr. Ayhan ŞAHİN,

Department of Anesthesiology and Reanimation, Medical Faculty of Namık Kemal University, Tekirdağ, Turkey

Namık Kemal University Medicine Faculty, Anesthesiology Department, 2nd Floor, Tekirdağ, Süleymanpaşa, 59100, Turkey

**Phone number:** 0905324730503

E-mail: drayhan.sahin@hotmail.com

Co-authors: Ahmet GÜLTEKİN1, Gülcan GÜCER ŞAHİN2, İlker YILDIRIM1, Onur BARAN1, Tolga ERSÖZ3, M.Cavidan ARAR1

1Department of Anesthesiology and Reanimation, Medical Faculty of Namık Kemal University, Tekirdağ, Turkey

2Department of Radiology, Medical Faculty of Namık Kemal University, Tekirdağ, Turkey 3Department of Otolaryngology, Medical Faculty of Namık Kemal University, Tekirdağ, Turkey

## Statistical analysis

Descriptive statistics were given as mean  $\pm$  standard deviation and median with interquartile range (IQR) of 25% to 75% for continuous variables depending on their distribution. Numbers and percentages were used for categorical variables. The numerical variables' normal distribution was analyzed by the Kolmogorov-Smirnov test and checked by Q-Q plots and histograms. The Levene test checked the homogeneity of the variances.

In comparing two independent groups, the Independent Samples t-test was used where numerical variables had a normal distribution. For variables without normal distribution, the Mann-Whitney U test was applied.

To compare the differences between categorical variables, Pearson Chi-Square and Fisher's Exact tests were used in 2x2 tables. For comparison of differences between categorical variables, Fisher Freeman Halton test was used in RxC tables.

For statistical analysis, "Jamovi project (2020), Jamovi (Version 1.6.8) [Computer Software] (Retrieved from https://www.jamovi.org), and JASP (Version 0.14) (Retrieved from https://jasp-stats.org) were used. The significance level (p-value) was set at 0.05 in all statistical analyses.

Forty-two subjects were screened for eligibility from June 2020 to December 2020. Eleven patients did not meet inclusion criteria, and two patients declined to participate. After

informed consent, 29 patients were enrolled and randomized. There were no differences in subject characteristics between groups.

The study groups included 29 patients with a mean age of  $62.66 \pm 13.25$  years. There were 14 (48.3%) and 15 patients (51.7%) in Group S and Group ST. The majority of the patients (70.0%) were male. Larynx cancer was the most frequent diagnosis (70.0%) in the study groups. The groups were similar regarding age, sex distribution, and pathological diagnoses.